CLINICAL TRIAL: NCT00529256
Title: Evaluation of Organisational Changes to Promote Smoking Cessation
Acronym: ESCMMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Lakes Research Into Practice Network (Network)
Collaborators: Robert Wood Johnson Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 61-6498
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Last update posted 2007-09-14 (Estimated); Status verified 2005-04

CONDITIONS: Adult Smokers
Keywords: Adult smokers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (No Intervention): No intervention
  Interventions: Behavioral: Feeback group

INTERVENTIONS:
Behavioral: Feeback group — The intervention practices received a quarterly comparative feedback performance report based on the Achievable Benchmarks of Care (ABC) research conducted by Kieffe (YEAR).

SUMMARY:
The Department of Family Practice at Michigan State University partnered with BCBSM with a grant from the Robert Wood Johnson Foundation to recruit primary care practices for a 3 year study designed to assess smoking cessation referral rates by primary care physicians in Michigan.

DETAILED DESCRIPTION:
There are two main research questions to our study: 1) Whether provider referral rates to smoking cessation services and quitline counseling are enhanced by comparative feedback profiles to individual providers and provider groups (Study 1) and 2) Whether health plan members who receive pharmacotherapy for smoking cessation have higher participation rates in smoking cessation services if they receive proactive, invitational phone calls (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* Primary care practice and thier Adult smokers

Exclusion Criteria:

* Non somkers

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2001-12; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
evaluate and provide a model of smoking cessation interventions

CONTACTS AND LOCATIONS:
Overall Officials: William Wadland, MD, MS, Principal Investigator — Michigan State University
Locations (1):
- William Wadland, East Lansing, Michigan, United States

REFERENCES:
- [Derived] Holtrop JS, Malouin R, Weismantel D, Wadland WC. Clinician perceptions of factors influencing referrals to a smoking cessation program. BMC Fam Pract. 2008 Mar 28;9:18. doi: 10.1186/1471-2296-9-18. PMID 18373854